CLINICAL TRIAL: NCT03541109
Title: Fixed Combination Therapy for Secondary Prevention of Major Cardiovascular Events
Brief Title: A Polypill for Secondary Prevention of Ischemic Heart Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoumeh Sadeghi, Head of Cardiac Rehabilitation Research Center, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Persian Polypill
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Acute Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction
Keywords: Cardiovascular disease; fixed dose combination therapy; cost effectiveness
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polypill (Experimental): Polypill group will receive a fixed dose combinations of aspirin (81mg), atorvastatin (40mg), metoprolol (50 mg), and Valsartan (40 mg), prescribed once daily by moth for 34 months
  Interventions: Drug: Polypill
- Control (No Intervention): The usual care arm will receive regular drug order at the time of discharge from the hospital.

INTERVENTIONS:
Drug: Polypill — fixed dose combination of aspirin (81mg), atorvastatin (40mg), metoprolol (50 mg), and Valsartan (40 mg)
  Other Names: Polypill-S
  Arms: Polypill

SUMMARY:
Cardiovascular diseases (CVD) are the leading cause of mortality and morbidity worldwide. The most important aspect of CVD secondary prevention is adherence to guideline-indicated pharmacological therapy which globally remains low. In previous studies, a Polypill containing fixed dose combination of essential drugs have improved patient adherence to these drugs. The effect of such a strategy on pharmacological therapy uptake, cost-effectiveness, and CVD recurrence in our setting will be assessed in this study. Participants hospitalized in three referral hospitals in Isfahan, Iran because of an acute myocardial infarction (MI) (ST elevation MI (STEMI) or non-ST elevation MI (NSTEMI)) will be randomized to either receiving Polypill or usual care after MI. Patient recruitment will be carried out at the time of patient discharge from the hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized because of an acute myocardial infarction (STEMI/NSTEMI) and alive after discharge for at least 1 month
* signing informed consent
* clear indication of receiving all components of Polypill (aspirin, statin, ACE inhibitor/ARB, and beta blocker)
* living in Isfahan city or nearby areas so that they can attend follow-ups
* No mental illness limiting their self-care ability or Severe illness with an estimated lifespan of less than 3 years
* No history of adverse reaction or contraindication to any component of the Polypill
* Not having Secondary hyperlipidemia, serum creatinine ≥ 2, severe heart failure
* No plan for a procedure (CABG, PCI, or another surgical procedures) within following 6 months

Exclusion Criteria:

* Patient unlikely to complete trial
* Need to change or discontinue any of the four principal drugs of the Polypill to achieve better control of the disease or risk factors or because of adverse drug reactions (based on physician's idea)
* Severe illness with an estimated lifespan of less than 3 years

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
A composite clinical outcome of major adverse cardiovascular events (MACE) | from time of randomization up to 34 months
  MACE includes cardiac death, fatal/nonfatal MI or stroke, hospitalization due to acute coronary syndrome/acute cerebrovascular accident, revascularization procedures, development or worsening of HF, and development of persistent new AF.

SECONDARY OUTCOMES:
cost-effectiveness of Polypill treatment compared with usual care | up to 34 months
  The analysis will be done on direct and indirect costs of treatment. Direct costs will be assessed from perspective of health care system. Current Iranian public medical tariffs will be the base of calculations. The incremental cost effectiveness ratio (ICER) will be calculated for primary outcomes.

OTHER OUTCOMES:
drug related adverse events | 1 month
  assessed by a questionnaire filled by the responsible physician
drug related adverse events | 4 months
  assessed by a questionnaire filled by the responsible physician
drug related adverse events | 10 months
  assessed by a questionnaire filled by the responsible physician
drug related adverse events | 22 months
  assessed by a questionnaire filled by the responsible physician
drug related adverse events | 34 months
  assessed by a questionnaire filled by the responsible physician
patient satisfaction with drug consumption | 1 month
  Satisfaction Questionnaire for Medication (TSQM)
patient satisfaction with drug consumption | 4 months
  Satisfaction Questionnaire for Medication (TSQM)
patient satisfaction with drug consumption | 10 months
  Satisfaction Questionnaire for Medication (TSQM)
patient satisfaction with drug consumption | 22 months
  Satisfaction Questionnaire for Medication (TSQM)
patient satisfaction with drug consumption | 34 months
  Satisfaction Questionnaire for Medication (TSQM)
health related quality of life | 1 month
  Validated Persian version of the EuroQol-5D (EQ-5D)
health related quality of life | 4 months
  Validated Persian version of the EuroQol-5D (EQ-5D)
health related quality of life | 10 months
  Validated Persian version of the EuroQol-5D (EQ-5D)
health related quality of life | 22 months
  Validated Persian version of the EuroQol-5D (EQ-5D)
health related quality of life | 34 months
  Validated Persian version of the EuroQol-5D (EQ-5D)
changes in systolic blood pressure from baseline | baseline and 1 month
  average readings of systolic blood pressure measured two times (at least 3 min apart) at sitting position
changes in systolic blood pressure from baseline | baseline and 4 months
  average readings of systolic blood pressure measured two times (at least 3 min apart) at sitting position
changes in systolic blood pressure from baseline | baseline and 10 months
  average readings of systolic blood pressure measured two times (at least 3 min apart) at sitting position
changes in systolic blood pressure from baseline | baseline and 22 months
  average readings of systolic blood pressure measured two times (at least 3 min apart) at sitting position
changes in systolic blood pressure from baseline | baseline and 34 months
  average readings of systolic blood pressure measured two times (at least 3 min apart) at sitting position
change in serum LDL from baseline | baseline and 1 month
  fasting Low Density Lipoprotein Cholesterol (LDL-C)
change in serum LDL from baseline | baseline and 4 months
  fasting Low Density Lipoprotein Cholesterol (LDL-C)
change in serum LDL from baseline | baseline and 10 months
  fasting Low Density Lipoprotein Cholesterol (LDL-C)
change in serum LDL from baseline | baseline and 22 months
  fasting Low Density Lipoprotein Cholesterol (LDL-C)
change in serum LDL from baseline | baseline and 34 months
  fasting Low Density Lipoprotein Cholesterol (LDL-C)
patient adherence to Aspirin at the final visit | 34 months
  patient is adherent if achieves a score of more than 6 from validated Persian version of Morisky-Medication Adherence Scale (8 item) Questionnaire (MMAS-8) (score: 0 to 8) and more than 85% of pills prescribed over last 3 months are consumed (pill count method)
patient adherence to Atorvastatin at the final visit | 34 months
  MMAS-8 questionnaire and pill count
patient adherence to Metoprolol at the final visit | 34 months
  MMAS-8 questionnaire and pill count
patient adherence to valsartan at the final visit | 34 months
  MMAS-8 questionnaire and pill count
patient adherence to Aspirin, Atorvastatin, Metoprolol, Valsartan | 1 month
  MMAS-8 questionnaire and pill count
patient adherence to Aspirin, Atorvastatin, Metoprolol, Valsartan | 4 months
  MMAS-8 questionnaire and pill count
patient adherence to Aspirin, Atorvastatin, Metoprolol, Valsartan | 10 months
  MMAS-8 questionnaire and pill count
patient adherence to Aspirin, Atorvastatin, Metoprolol, Valsartan | 22 months
  MMAS-8 questionnaire and pill count

CONTACTS AND LOCATIONS:
Overall Officials: Masoumeh Sadeghi, professor, Principal Investigator — Isfahan Cardiovascular Research Center, Cardiovascular Research Institute, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (2):
- Iran (2):
  - Chamran cardiology hospital, Isfahan
  - Cardiovascular Research Institute, Isfahan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after study completion
Access Criteria: Requests will be assessed by a responsible panel after signing a data access agrement.
URL: http://icri.mui.ac.ir/